CLINICAL TRIAL: NCT04972526
Title: Evaluation of the Clinical Impact and Safety of Focused Transesophageal Echocardiography During Resuscitation of Critically Ill Patients in the Emergency Department and Intensive Care Settings
Brief Title: Resuscitative TEE Collaborative Registry
Acronym: rTEECoRe
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Felipe Teran, MD, MSCE, Chair, Resuscitative TEE Collaborative Registry, Weill Medical College of Cornell University
Other Study IDs: 844522
Record Dates: First submitted 2021-06-15; First posted 2021-07-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Arrest; Cardiac Arrest Circulatory; Cardiac Arrest, Out-Of-Hospital; Shock; Hemodynamic Instability
Keywords: Transesophageal Echocardiography; Resuscitation; Cardiac Arrest; Point-of-care Ultrasound; Focused Cardiac Ultrasound
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Out-of-hospital Cardiac Arrest: Patients receiving TEE as part of their clinical evaluation during cardiac arrest that occurred outside the hospital (e.g. in/at a home or residence, in a public area, during transport to the emergency department, etc.)
- In-hospital Cardiac Arrest: Patients receiving TEE as part of the clinical evaluation during cardiac arrest that occurred within a hospital (e.g in the emergency department, an Intensive Care Unit, a hospital ward, the operating room, etc.)
- Undifferentiated Shock or Acute Hemodynamic Decompensation: Patients receiving TEE as part of the initial evaluation of undifferentiated shock or acute hemodynamic decompensation
- Hemodynamic Monitoring in a Critically Ill Patient: Critically ill patients receiving TEE as part of hemodynamic monitoring
- Procedural Guidance: Patients receiving TEE as a means to assist providers performing procedures (e.g. intravenous pacemaker placement, veno-arterial or veno-venous extracorporeal membrane oxygenation [ECMO], impella heart pump placement, intra-aortic balloon pump placement, etc.)

SUMMARY:
The general objective of this study is to evaluate the clinical impact and safety of focused, point-of-care transesophageal echocardiography (TEE) used during the evaluation of critically-ill patients in the emergency and intensive care settings. The target population for this study are critically-ill patients over the age of 18 who as part of their routine clinical care are receiving a focused TEE.

The primary objective of this study is to determine the clinical impact and safety of TEE performed during the evaluation of critically-ill patients in the emergency department and intensive care settings.

The secondary objective(s) of this study are to characterize the use of this imaging modality in the subsets of critically-ill patients in shock and cardiac arrest; including but not limited to; description of the frequency of studies, clinical indications, clinician characteristics, echocardiography findings, timing of studies, procedure-related complications and patient outcomes.

DETAILED DESCRIPTION:
Vision

The Resuscitative TEE Collaborative Registry aims to accelerate the development of outcome-oriented research and knowledge translation on the use of TEE in emergency and critical care settings.

Mission

The registry aims to catalyze clinical research involving the use of TEE in critically-ill patients through the following strategic initiatives:

* Facilitate collaboration between different clinical teams and organizations across the entire spectrum of users of TEE in acute care setting, including emergency departments and intensive care units.
* Standardize data collection and reporting that enables multi-institutional data sharing.
* Provide an efficient research infrastructure that facilitates data capture, management and analysis, enabling teams around the world to conduct research studies in this field.
* Make shared data open and accessible to clinicians and researchers.

ELIGIBILITY:
Inclusion Criteria:

* Adult critically-ill patients who as part of their routine clinical care receive focused TEE in the emergency department of intensive care setting.

Exclusion Criteria:

* Children (age under 18 years)
* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically-ill patients who as part of their routine clinical care receive focused TEE in the emergency department of intensive care setting.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
The clinical impact and safety of TEE performed during the evaluation of critically ill patients in the emergency department and intensive care settings. | From the time of admission to the hospital until the date of discharge from the hospital or date of death from any cause, whichever occurs first, assessed up to 12 weeks
  Determination of ROSC and survival to hospital discharge

SECONDARY OUTCOMES:
The use of the TEE imaging modality in subsets of critically-ill patients in shock and cardiac arrest. | From the time of admission to the hospital until the date of discharge from the hospital or date of death from any cause, whichever occurs first, assessed up to 12 weeks
  Description of the frequency of studies, clinical indications, clinician characteristics, echocardiography findings, timing of studies, procedure-related complications and patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Teran, MD, MSCE, Principal Investigator — Weill Medical College of Cornell University; Clark G Owyang, MD, Study Chair — Weill Medical College of Cornell University
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
After the first year the registry gathers data, investigators from participating centers will have the opportunity to propose studies and request data pertaining to specific study aims.

REFERENCES:
- [Background] Teran F, Prats MI, Nelson BP, Kessler R, Blaivas M, Peberdy MA, Shillcutt SK, Arntfield RT, Bahner D. Focused Transesophageal Echocardiography During Cardiac Arrest Resuscitation: JACC Review Topic of the Week. J Am Coll Cardiol. 2020 Aug 11;76(6):745-754. doi: 10.1016/j.jacc.2020.05.074. PMID 32762909
- [Background] Teran F, Burns KM, Narasimhan M, Goffi A, Mohabir P, Horowitz JM, Yuriditsky E, Nagdev A, Panebianco N, Chin EJ, Gottlieb M, Koenig S, Arntfield R. Critical Care Transesophageal Echocardiography in Patients during the COVID-19 Pandemic. J Am Soc Echocardiogr. 2020 Aug;33(8):1040-1047. doi: 10.1016/j.echo.2020.05.022. Epub 2020 May 23. PMID 32600742
- [Background] Teran F, Dean AJ, Centeno C, Panebianco NL, Zeidan AJ, Chan W, Abella BS. Evaluation of out-of-hospital cardiac arrest using transesophageal echocardiography in the emergency department. Resuscitation. 2019 Apr;137:140-147. doi: 10.1016/j.resuscitation.2019.02.013. Epub 2019 Feb 16. PMID 30779977
- [Background] Arntfield R, Lau V, Landry Y, Priestap F, Ball I. Impact of Critical Care Transesophageal Echocardiography in Medical-Surgical ICU Patients: Characteristics and Results From 274 Consecutive Examinations. J Intensive Care Med. 2020 Sep;35(9):896-902. doi: 10.1177/0885066618797271. Epub 2018 Sep 6. PMID 30189783
- [Background] Lerner RP, Haaland A, Lin J. Temporary transvenous pacer placement under transesophageal echocardiogram guidance in the Emergency Department. Am J Emerg Med. 2020 May;38(5):1044.e3-1044.e4. doi: 10.1016/j.ajem.2019.12.027. Epub 2019 Dec 16. PMID 31870671
- [Background] Catena E, Ottolina D, Fossali T, Rech R, Borghi B, Perotti A, Ballone E, Bergomi P, Corona A, Castelli A, Colombo R. Association between left ventricular outflow tract opening and successful resuscitation after cardiac arrest. Resuscitation. 2019 May;138:8-14. doi: 10.1016/j.resuscitation.2019.02.027. Epub 2019 Feb 27. PMID 30825552
- [Background] Osman A, Fong CP, Wahab SFA, Panebianco N, Teran F. Transesophageal Echocardiography at the Golden Hour: Identification of Blunt Traumatic Aortic Injuries in the Emergency Department. J Emerg Med. 2020 Sep;59(3):418-423. doi: 10.1016/j.jemermed.2020.05.003. Epub 2020 Jun 23. PMID 32591302
- [Background] Hwang SO, Zhao PG, Choi HJ, Park KH, Cha KC, Park SM, Kim SC, Kim H, Lee KH. Compression of the left ventricular outflow tract during cardiopulmonary resuscitation. Acad Emerg Med. 2009 Oct;16(10):928-33. doi: 10.1111/j.1553-2712.2009.00497.x. Epub 2009 Sep 3. PMID 19732038
- [Background] Fair J 3rd, Mallin MP, Adler A, Ockerse P, Steenblik J, Tonna J, Youngquist ST. Transesophageal Echocardiography During Cardiopulmonary Resuscitation Is Associated With Shorter Compression Pauses Compared With Transthoracic Echocardiography. Ann Emerg Med. 2019 Jun;73(6):610-616. doi: 10.1016/j.annemergmed.2019.01.018. Epub 2019 Feb 14. PMID 30773413
- [Background] Parker BK, Salerno A, Euerle BD. The Use of Transesophageal Echocardiography During Cardiac Arrest Resuscitation: A Literature Review. J Ultrasound Med. 2019 May;38(5):1141-1151. doi: 10.1002/jum.14794. Epub 2018 Oct 2. PMID 30280396
- [Background] Teran F. Resuscitative Cardiopulmonary Ultrasound and Transesophageal Echocardiography in the Emergency Department. Emerg Med Clin North Am. 2019 Aug;37(3):409-430. doi: 10.1016/j.emc.2019.03.003. Epub 2019 May 21. PMID 31262412
- [Background] Jaidka A, Hobbs H, Koenig S, Millington SJ, Arntfield RT. Better With Ultrasound: Transesophageal Echocardiography. Chest. 2019 Jan;155(1):194-201. doi: 10.1016/j.chest.2018.09.023. Epub 2018 Oct 9. PMID 30312590
- [Background] Vieillard-Baron A, Chergui K, Rabiller A, Peyrouset O, Page B, Beauchet A, Jardin F. Superior vena caval collapsibility as a gauge of volume status in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1734-9. doi: 10.1007/s00134-004-2361-y. Epub 2004 Jun 26. PMID 15375649
- [Background] Blaivas M. Transesophageal echocardiography during cardiopulmonary arrest in the emergency department. Resuscitation. 2008 Aug;78(2):135-40. doi: 10.1016/j.resuscitation.2008.02.021. Epub 2008 May 16. PMID 18486300
- [Background] Arntfield R, Pace J, McLeod S, Granton J, Hegazy A, Lingard L. Focused transesophageal echocardiography for emergency physicians-description and results from simulation training of a structured four-view examination. Crit Ultrasound J. 2015 Dec;7(1):27. doi: 10.1186/s13089-015-0027-3. Epub 2015 Jun 12. PMID 26123608
- [Background] Arntfield R, Pace J, Hewak M, Thompson D. Focused Transesophageal Echocardiography by Emergency Physicians is Feasible and Clinically Influential: Observational Results from a Novel Ultrasound Program. J Emerg Med. 2016 Feb;50(2):286-94. doi: 10.1016/j.jemermed.2015.09.018. Epub 2015 Oct 24. PMID 26508495
- [Background] Fair J, Tonna J, Ockerse P, Galovic B, Youngquist S, McKellar SH, Mallin M. Emergency physician-performed transesophageal echocardiography for extracorporeal life support vascular cannula placement. Am J Emerg Med. 2016 Aug;34(8):1637-9. doi: 10.1016/j.ajem.2016.06.038. Epub 2016 Jun 7. PMID 27318746
- [Background] Byars DV, Tozer J, Joyce JM, Vitto MJ, Taylor L, Kayagil T, Jones M, Bishop M, Knapp B, Evans D. Emergency Physician-performed Transesophageal Echocardiography in Simulated Cardiac Arrest. West J Emerg Med. 2017 Aug;18(5):830-834. doi: 10.5811/westjem.2017.5.33543. Epub 2017 Jul 19. PMID 28874934
- [Background] Fair J, Mallin M, Mallemat H, Zimmerman J, Arntfield R, Kessler R, Bailitz J, Blaivas M. Transesophageal Echocardiography: Guidelines for Point-of-Care Applications in Cardiac Arrest Resuscitation. Ann Emerg Med. 2018 Feb;71(2):201-207. doi: 10.1016/j.annemergmed.2017.09.003. Epub 2017 Nov 6. PMID 29107407
- See also: Registry Home at the Center for Resuscitation Science — https://www.med.upenn.edu/resuscitation/rteecore/
- See also: Resuscitative TEE Project Home — https://www.resuscitativetee.com

DOCUMENTS (1):
  • Study Protocol (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04972526/Prot_000.pdf